CLINICAL TRIAL: NCT06865274
Title: Multicenter Prospective Interventional Study to Evaluate the Frequency of FCGR3A Gene Polymorphisms in Patients With Neuromyelitis Optica Spectrum Disorders, Myelin Oligodendrocyte Glycoprotein Antibody Disease, and Multiple Sclerosis.
Brief Title: Frequency of FCGR3A Gene Polymorphisms in Patients With Neuromyelitis Optica Spectrum Disorders, Anti-oligodendrocyte Myelin Protein Antibody Disease, and Multiple Sclerosis.
Acronym: PoGe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mirabella Massimiliano, Associate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 7168
Record Dates: First submitted 2025-02-21; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Neuromyelitis Optica Spectrum Disorders; MOGAD; Multiple Sclerosis
Keywords: NMOSD; MOGAD; MS; polymorphysm; FCG3A
MeSH Terms: conditions — Neuromyelitis Optica; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients diagnosied with neuromyelitis optica spectrum disorder and MOG antibodies associated diseas (Other): Patients will undergo a peripheral venous blood draw of approximately 5 ml (collected in EDTA) during routine blood tests for DNA extraction and genetic analysis, limited to the reserach of FCG3A polymorphisms. The results obtained will be compared with a control-group composed by patients diagnosed with Multiple sclerosis.
  Interventions: Procedure: Blood draw for the laboratory assessment
- Patients diagnosied with Multiple Sclerosis (Other): Patients will undergo a peripheral venous blood draw of approximately 5 ml (collected in EDTA) during routine blood tests for DNA extraction and genetic analysis, limited to the reserach of FCG3A polymorphisms. This is a comparison group.
  Interventions: Procedure: Blood draw for the laboratory assessment

INTERVENTIONS:
Procedure: Blood draw for the laboratory assessment — Blood draw of approximately 5 ml of peripheral venous blood (collected in EDTA) will be collected for DNA extraction and genetic analysis limited to the research of FCG3A polymorphisms

SUMMARY:
The goal of this study is to assess the frequency of genetic polymorphisms of the FCG3A in a cohort of Italian patients affected by neuromyelitis optica spectrum disorder (NMOSD) and mog antibody associated disease (MOGAD) and in a a comparison group of patients affected with Multiple Sclerosis (MS).

The study will involve adult patients diagnosed with MS, NMOSD, or MOGAD, followed at various clinical centers in the Lazio region.

Patients from the participating clinical centers will be selected, and their medical records will be analyzed to collect clinical and neuroimaging data. The data will include demographic information such as age, sex and body mass index and clinical information such as age at disease onset, disease duration, antibody status (AQP4+/- and MOG+/-), disease-modifying therapies, as well as MRI data and the Expanded Disability Status Scale (EDSS) score.

Each patient included in the study will undergo a single blood draw of approximately 5 ml of peripheral venous blood during routine blood tests, which will be used for DNA extraction and polimorphysm analysis. Demographic and clinical differences between patients with NMOSD and MOGAD, with and without the polymorphism, will be assessed and compared with the group of patients with MS.

DETAILED DESCRIPTION:
FCG receptors (FCGR) are proteins expressed by various immune cells that bind to the Fc portion of immunoglobulin G (IgG). They play a key role in innate and adaptive immunity, regulating inflammatory responses and preventing autoimmunity. Genetic studies have shown that variations in FCGR genes can influence these functions, altering phagocytosis capacity and inflammatory response.

One particularly relevant polymorphism is SNP rs396991 in the FCGR3A gene, which encodes the receptor expressed on NK cells, monocytes, and macrophages. This SNP causes the substitution of the amino acid phenylalanine (F) with valine (V) at position 158, modifying the receptor's affinity for IgG. The 158V variant is associated with an enhanced inflammatory response, while 158F is linked to reduced immune complex clearance, contributing to the pathogenesis of autoimmune diseases such as lupus, rheumatoid arthritis, and sarcoidosis.

Neuromyelitis optica spectrum disorder (NMOSD) and myelin oligodendrocyte glycoprotein antibody-associated disease (MOGAD) are two inflammatory disorders of the central nervous system, often severe and recurrent. NMOSD is characterized by autoantibodies against aquaporin-4 (AQP4), while MOGAD is associated with autoantibodies against MOG glycoprotein. There are currently no data on the frequency of the rs396991 polymorphism in the Italian population affected by these diseases.

The primary objective of this study is to assess the frequency of the FCGR3A-V158F genetic polymorphism in a cohort of Italian patients affected by NMOSD and MOGAD. A comparison group composed of patients diagnosed with Multiple Sclerosis (MS) will also be included.

The study will involve adult patients diagnosed with MS, NMOSD, or MOGAD, receiving care at various clinical centers in the Lazio region. Patients from the participating clinical centers will be selected, and their medical records, both paper-based and digital, will be reviewed to collect clinical and neuroimaging data. These data will be organized in an Excel database and will include information such as age, sex, ethnic background, body mass index, smoking status, presence of other autoimmune diseases, and non-neurological comorbidities. Additional recorded information will include diagnosis (NMOSD, MS, or MOGAD), age at disease onset, disease duration, antibody status (AQP4+/- and MOG+/-), previous disease-modifying therapies and their duration, as well as MRI data and Expanded Disability Status Scale (EDSS) scores.

For genetic analysis, each patient included in the study will undergo a blood draw of approximately 5 ml of peripheral venous blood (collected in EDTA) during routine blood tests. The sample will be used for DNA extraction, following the patient's signed informed consent. Genetic investigations will be conducted at the Genomic Medicine Section of the Department of Life Sciences and Public Health at Università Cattolica del Sacro Cuore in Rome. DNA samples will be stored anonymously for up to 10 years from the start of the project, with access restricted to authorized personnel. Patients or their families may request the destruction of their DNA at any time.

A total of 50 patients will be recruited, with a 12-month enrollment period and a total study duration of 24 months. The secondary objective is to identify potential differences in the clinical characteristics of NMOSD and MOGAD patients who express the polymorphism compared to those who do not.

Genetic analyses will be conducted at the Section of Genomic Medicine, Department of Life Sciences and Public Health, Università Cattolica del Sacro Cuore (Rome). The extracted DNA will be stored anonymously with an alphanumeric code for a maximum of 10 years from the start date of the project at the same institution. Only a limited number of authorized personnel will have access to the samples and data, subject to approval from the principal investigator (Prof. Massimiliano Mirabella). If requested by the patient or their family, the DNA can be destroyed at any time.

DNA extraction will be performed using the Wizard Genomic DNA Isolation Kit (Promega) and quantified via spectrophotometer (Thermo Fisher) and agarose gel electrophoresis. The detection of the rs396991 polymorphism in the FCGR3A gene in patients with NMOSD, MS, and MOGAD will be carried out using Sanger sequencing, employing primers described by Mahaweni et al. (14).

The presence of Copy Number Variable Regions (CNRs) in the FCGR3A gene will be assessed through MLPA (MRC Holland) and will be reserved only for patients who test negative for the rs396991 polymorphism using the Sanger method.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with MS, NMOSD, or MOGAD receiving care at participating centers
* Patients aged ≥ 18 years
* Ability to understand and sign informed consent

Exclusion Criteria:

* Individuals under 18 years of age
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
FCGR3A gene polymorphism frequency in a cohort of Italian patients affected by NMOSD and MOGAD. | Baseline
  To assess the frequency of the FCGR3A gene polymorphism in a cohort of Italian patients affected by NMOSD and MOGAD.

SECONDARY OUTCOMES:
Clinical characteristics of NMOSD and MOGAD patients who express the polymorphism | From enrollment to 24 months
  Disability assessed by Expanded disability status scale in NMOSD and MOGAD patients who express the polymorphism and in to those who do not.
Clinical characteristics of NMOSD and MOGAD patients who express the polymorphism | From enrollment to 24 months
  Number of disease relapses in patients with NMOSD and MOGAD expressing the polymorphisms and in patients without the polymorphism

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodin DS. The epidemiology of multiple sclerosis: insights to disease pathogenesis. Handb Clin Neurol. 2014;122:231-66. doi: 10.1016/B978-0-444-52001-2.00010-8. PMID 24507521
- [Background] Jakimovski D, Bittner S, Zivadinov R, Morrow SA, Benedict RH, Zipp F, Weinstock-Guttman B. Multiple sclerosis. Lancet. 2024 Jan 13;403(10422):183-202. doi: 10.1016/S0140-6736(23)01473-3. Epub 2023 Nov 7. PMID 37949093
- [Background] Banwell B, Bennett JL, Marignier R, Kim HJ, Brilot F, Flanagan EP, Ramanathan S, Waters P, Tenembaum S, Graves JS, Chitnis T, Brandt AU, Hemingway C, Neuteboom R, Pandit L, Reindl M, Saiz A, Sato DK, Rostasy K, Paul F, Pittock SJ, Fujihara K, Palace J. Diagnosis of myelin oligodendrocyte glycoprotein antibody-associated disease: International MOGAD Panel proposed criteria. Lancet Neurol. 2023 Mar;22(3):268-282. doi: 10.1016/S1474-4422(22)00431-8. Epub 2023 Jan 24. PMID 36706773
- [Background] Wingerchuk DM, Lucchinetti CF. Neuromyelitis Optica Spectrum Disorder. N Engl J Med. 2022 Aug 18;387(7):631-639. doi: 10.1056/NEJMra1904655. No abstract available. PMID 36070711
- [Background] Whittam DH, Tallantyre EC, Jolles S, Huda S, Moots RJ, Kim HJ, Robertson NP, Cree BAC, Jacob A. Rituximab in neurological disease: principles, evidence and practice. Pract Neurol. 2019 Feb;19(1):5-20. doi: 10.1136/practneurol-2018-001899. Epub 2018 Nov 29. PMID 30498056
- [Background] Manger K, Repp R, Jansen M, Geisselbrecht M, Wassmuth R, Westerdaal NA, Pfahlberg A, Manger B, Kalden JR, van de Winkel JG. Fcgamma receptor IIa, IIIa, and IIIb polymorphisms in German patients with systemic lupus erythematosus: association with clinical symptoms. Ann Rheum Dis. 2002 Sep;61(9):786-92. doi: 10.1136/ard.61.9.786. PMID 12176802
- [Background] Dijstelbloem HM, Scheepers RH, Oost WW, Stegeman CA, van der Pol WL, Sluiter WJ, Kallenberg CG, van de Winkel JG, Tervaert JW. Fcgamma receptor polymorphisms in Wegener's granulomatosis: risk factors for disease relapse. Arthritis Rheum. 1999 Sep;42(9):1823-7. doi: 10.1002/1529-0131(199909)42:93.0.CO;2-X. PMID 10513795
- [Background] Capiod T. Cell proliferation, calcium influx and calcium channels. Biochimie. 2011 Dec;93(12):2075-9. doi: 10.1016/j.biochi.2011.07.015. Epub 2011 Jul 23. PMID 21802482
- [Background] Iannuzzi MC, Iyengar SK, Gray-McGuire C, Elston RC, Baughman RP, Donohue JF, Hirst K, Judson MA, Kavuru MS, Maliarik MJ, Moller DR, Newman LS, Rabin DL, Rose CS, Rossman MD, Teirstein AS, Rybicki BA. Genome-wide search for sarcoidosis susceptibility genes in African Americans. Genes Immun. 2005 Sep;6(6):509-18. doi: 10.1038/sj.gene.6364235. PMID 15951742
- [Background] Chen JY, Wang CM, Tsao KC, Chow YH, Wu JM, Li CL, Ho HH, Wu YJ, Luo SF. Fcgamma receptor IIa, IIIa, and IIIb polymorphisms of systemic lupus erythematosus in Taiwan. Ann Rheum Dis. 2004 Jul;63(7):877-80. doi: 10.1136/ard.2003.005892. PMID 15194589
- [Background] Morgan AW, Griffiths B, Ponchel F, Montague BM, Ali M, Gardner PP, Gooi HC, Situnayake RD, Markham AF, Emery P, Isaacs JD. Fcgamma receptor type IIIA is associated with rheumatoid arthritis in two distinct ethnic groups. Arthritis Rheum. 2000 Oct;43(10):2328-34. doi: 10.1002/1529-0131(200010)43:103.0.CO;2-Z. PMID 11037893
- [Background] Typiak MJ, Rebala K, Dudziak M, Dubaniewicz A. Polymorphism of FCGR3A gene in sarcoidosis. Hum Immunol. 2014 Apr;75(4):283-8. doi: 10.1016/j.humimm.2014.02.011. Epub 2014 Feb 12. PMID 24530756
- [Background] Asano K, Matsumoto T, Umeno J, Hirano A, Esaki M, Hosono N, Matsui T, Kiyohara Y, Nakamura Y, Kubo M, Kitazono T. Impact of allele copy number of polymorphisms in FCGR3A and FCGR3B genes on susceptibility to ulcerative colitis. Inflamm Bowel Dis. 2013 Sep;19(10):2061-8. doi: 10.1097/MIB.0b013e318298118e. PMID 23917248
- [Background] Nieto A, Caliz R, Pascual M, Mataran L, Garcia S, Martin J. Involvement of Fcgamma receptor IIIA genotypes in susceptibility to rheumatoid arthritis. Arthritis Rheum. 2000 Apr;43(4):735-9. doi: 10.1002/1529-0131(200004)43:43.0.CO;2-Q. PMID 10765917
- [Background] Edberg JC, Langefeld CD, Wu J, Moser KL, Kaufman KM, Kelly J, Bansal V, Brown WM, Salmon JE, Rich SS, Harley JB, Kimberly RP. Genetic linkage and association of Fcgamma receptor IIIA (CD16A) on chromosome 1q23 with human systemic lupus erythematosus. Arthritis Rheum. 2002 Aug;46(8):2132-40. doi: 10.1002/art.10438. PMID 12209518
- [Background] Morgan AW, Robinson JI, Barrett JH, Martin J, Walker A, Babbage SJ, Ollier WE, Gonzalez-Gay MA, Isaacs JD. Association of FCGR2A and FCGR2A-FCGR3A haplotypes with susceptibility to giant cell arteritis. Arthritis Res Ther. 2006;8(4):R109. doi: 10.1186/ar1996. PMID 16846526
- [Background] Wu J, Edberg JC, Redecha PB, Bansal V, Guyre PM, Coleman K, Salmon JE, Kimberly RP. A novel polymorphism of FcgammaRIIIa (CD16) alters receptor function and predisposes to autoimmune disease. J Clin Invest. 1997 Sep 1;100(5):1059-70. doi: 10.1172/JCI119616. PMID 9276722
- [Background] Breunis WB, van Mirre E, Geissler J, Laddach N, Wolbink G, van der Schoot E, de Haas M, de Boer M, Roos D, Kuijpers TW. Copy number variation at the FCGR locus includes FCGR3A, FCGR2C and FCGR3B but not FCGR2A and FCGR2B. Hum Mutat. 2009 May;30(5):E640-50. doi: 10.1002/humu.20997. PMID 19309690
- [Background] McGovern DP, Gardet A, Torkvist L, Goyette P, Essers J, Taylor KD, Neale BM, Ong RT, Lagace C, Li C, Green T, Stevens CR, Beauchamp C, Fleshner PR, Carlson M, D'Amato M, Halfvarson J, Hibberd ML, Lordal M, Padyukov L, Andriulli A, Colombo E, Latiano A, Palmieri O, Bernard EJ, Deslandres C, Hommes DW, de Jong DJ, Stokkers PC, Weersma RK; NIDDK IBD Genetics Consortium; Sharma Y, Silverberg MS, Cho JH, Wu J, Roeder K, Brant SR, Schumm LP, Duerr RH, Dubinsky MC, Glazer NL, Haritunians T, Ippoliti A, Melmed GY, Siscovick DS, Vasiliauskas EA, Targan SR, Annese V, Wijmenga C, Pettersson S, Rotter JI, Xavier RJ, Daly MJ, Rioux JD, Seielstad M. Genome-wide association identifies multiple ulcerative colitis susceptibility loci. Nat Genet. 2010 Apr;42(4):332-7. doi: 10.1038/ng.549. Epub 2010 Mar 14. PMID 20228799
- [Background] Yesmin K, Hargreaves C, Newby PR, Brand OJ, Heward JM, Franklyn JA, Gough SC, Simmonds MJ. Association of FcGRIIa with Graves' disease: a potential role for dysregulated autoantibody clearance in disease onset/progression. Clin Endocrinol (Oxf). 2010 Jul;73(1):119-25. doi: 10.1111/j.1365-2265.2010.03780.x. Epub 2010 Feb 10. PMID 20148910
- [Background] Khor CC, Davila S, Breunis WB, Lee YC, Shimizu C, Wright VJ, Yeung RS, Tan DE, Sim KS, Wang JJ, Wong TY, Pang J, Mitchell P, Cimaz R, Dahdah N, Cheung YF, Huang GY, Yang W, Park IS, Lee JK, Wu JY, Levin M, Burns JC, Burgner D, Kuijpers TW, Hibberd ML; Hong Kong-Shanghai Kawasaki Disease Genetics Consortium; Korean Kawasaki Disease Genetics Consortium; Taiwan Kawasaki Disease Genetics Consortium; International Kawasaki Disease Genetics Consortium; US Kawasaki Disease Genetics Consortium; Blue Mountains Eye Study. Genome-wide association study identifies FCGR2A as a susceptibility locus for Kawasaki disease. Nat Genet. 2011 Nov 13;43(12):1241-6. doi: 10.1038/ng.981. PMID 22081228
- [Background] Duan J, Lou J, Zhang Q, Ke J, Qi Y, Shen N, Zhu B, Zhong R, Wang Z, Liu L, Wu J, Wang W, Gong F, Miao X. A genetic variant rs1801274 in FCGR2A as a potential risk marker for Kawasaki disease: a case-control study and meta-analysis. PLoS One. 2014 Aug 5;9(8):e103329. doi: 10.1371/journal.pone.0103329. eCollection 2014. PMID 25093412
- [Background] Clark MR, Stuart SG, Kimberly RP, Ory PA, Goldstein IM. A single amino acid distinguishes the high-responder from the low-responder form of Fc receptor II on human monocytes. Eur J Immunol. 1991 Aug;21(8):1911-6. doi: 10.1002/eji.1830210820. PMID 1831131
- [Background] Warmerdam PA, van de Winkel JG, Vlug A, Westerdaal NA, Capel PJ. A single amino acid in the second Ig-like domain of the human Fc gamma receptor II is critical for human IgG2 binding. J Immunol. 1991 Aug 15;147(4):1338-43. PMID 1831223
- [Background] Willcocks LC, Carr EJ, Niederer HA, Rayner TF, Williams TN, Yang W, Scott JA, Urban BC, Peshu N, Vyse TJ, Lau YL, Lyons PA, Smith KG. A defunctioning polymorphism in FCGR2B is associated with protection against malaria but susceptibility to systemic lupus erythematosus. Proc Natl Acad Sci U S A. 2010 Apr 27;107(17):7881-5. doi: 10.1073/pnas.0915133107. Epub 2010 Apr 12. PMID 20385827
- [Background] Niederer HA, Willcocks LC, Rayner TF, Yang W, Lau YL, Williams TN, Scott JA, Urban BC, Peshu N, Dunstan SJ, Hien TT, Phu NH, Padyukov L, Gunnarsson I, Svenungsson E, Savage CO, Watts RA, Lyons PA, Clayton DG, Smith KG. Copy number, linkage disequilibrium and disease association in the FCGR locus. Hum Mol Genet. 2010 Aug 15;19(16):3282-94. doi: 10.1093/hmg/ddq216. Epub 2010 May 27. PMID 20508037
- [Background] Floto RA, Clatworthy MR, Heilbronn KR, Rosner DR, MacAry PA, Rankin A, Lehner PJ, Ouwehand WH, Allen JM, Watkins NA, Smith KG. Loss of function of a lupus-associated FcgammaRIIb polymorphism through exclusion from lipid rafts. Nat Med. 2005 Oct;11(10):1056-8. doi: 10.1038/nm1288. Epub 2005 Sep 18. PMID 16170323
- [Background] Nimmerjahn F, Ravetch JV. Fcgamma receptors as regulators of immune responses. Nat Rev Immunol. 2008 Jan;8(1):34-47. doi: 10.1038/nri2206. PMID 18064051
- [Background] Nimmerjahn F, Ravetch JV. FcgammaRs in health and disease. Curr Top Microbiol Immunol. 2011;350:105-25. doi: 10.1007/82_2010_86. PMID 20680807
- [Background] Bruhns P, Iannascoli B, England P, Mancardi DA, Fernandez N, Jorieux S, Daeron M. Specificity and affinity of human Fcgamma receptors and their polymorphic variants for human IgG subclasses. Blood. 2009 Apr 16;113(16):3716-25. doi: 10.1182/blood-2008-09-179754. Epub 2008 Nov 18. PMID 19018092